CLINICAL TRIAL: NCT07224321
Title: INHALE-1st: Technosphere Insulin (Afrezza®) In Combination With Basal Insulin For Youth With Newly-Diagnosed Type 1 Diabetes
Brief Title: INHALE-1st: Afrezza® For Youth With Newly-Diagnosed Type 1 Diabetes
Acronym: INHALE-1st
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-196
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus; Insulin; Inhaled; Afrezza; Technosphere; Pediatric; Inhaled Insulin; Type 1 Diabetes; Newly diagnosed type 1 diabetes; Technosphere Insulin; rapid-acting inhaled insulin; Meal-time inhaled insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance; Respiratory Aspiration | interventions — Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Afrezza (Technosphere Insulin) + Basal Insulin (Experimental): Individualized dose of Afrezza (Technosphere Insulin) and basal insulin for each patient before each meal (breakfast, lunch, and dinner) for 13 weeks.
  Interventions: Drug: Technosphere Insulin; Drug: Basal insulin

INTERVENTIONS:
Drug: Technosphere Insulin — 2 unit
  Other Names: Afrezza
Drug: Technosphere Insulin — 4, 8, 12 units
  Other Names: Afrezza
Drug: Basal insulin — subcutaneously-injected basal insulin

SUMMARY:
INHALE-1st is a Phase 2, single-arm, multi-center, clinical study evaluating the safety and efficacy of Afrezza in combination with subcutaneously-injected basal insulin (BI) for youth 10 to <18 years old with newly diagnosed stage 3 type 1 diabetes (T1D). The study will also evaluate the effect of an Afrezza plus BI reigmen on participant and parent/legally authorized representative satisfaction. Participants will be followed for 13 weeks during the main phase followed by an optional Extension Phase for participants continuing to use Afrezza in combination with BI for up to 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 to <18 years of age
* Clinical diagnosis of stage 3 T1D, per the investigator. Stage 3 is defined as hyperglycemia, meeting ADA glycemic and clinical diagnostic criteria
* Able to start the Afrezza-BI regimen within 10 days following T1D diagnosis (day 1 is based on the first insulin injection) if not hospitalized with diabetic ketoacidosis (DKA) and within 10 days of hospital discharge if hospitalized with DKA
* Forced Expiratory Volume in One Second (FEV1) >80.0% of predicted Global Lung Function Initiative (GLI) value
* Investigator believes that participant can be expected to follow the study protocol
* No medical, psychiatric, psychosocial conditions, or medications being taken that in the investigator's judgment would be a safety concern for participation in the study

Exclusion Criteria:

* Prior insulin treatment for stage 2 T1D
* History of chronic lung disease, such as asthma, or chronic obstructive pulmonary disease, lung cancer, or any other clinically important pulmonary disease (e.g., cystic fibrosis, bronchopulmonary dysplasia) in the judgment of the investigator
* Allergy or known hypersensitivity to human regular insulin
* Smoking (includes cigarettes, cigars, pipes, marijuana, and vaping devices) within 3 months prior to screening and/or positive cotinine test for smoking
* Positive urine pregnancy test for female subjects of childbearing potential

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Continuous Glucose Meter (CGM) measured time in range (TIR) ≥70% | 13 weeks
  Percentage of participants with a CGM-measured TIR 70-180 mg/dL ≥70% during 14 days prior to 13-week visit

SECONDARY OUTCOMES:
Mean Continuous Glucose Monitoring (CGM) glucose | 13 weeks
  Mean CGM glucose from baseline to 13 weeks
Continuous Glucose Monitoring (CGM) measured time-in-tight-range 70-140 mg/dL | 13 weeks
  Continuous Glucose Monitoring (CGM) measured time-in-tight-range 70-140 mg/dL from baseline to 13 weeks
Continuous Glucose Monitoring (CGM) measured percent time with glucose greater than 180 mg/dL | 13 weeks
  CGM-measured percent time with glucose > 180 mg/dL from baseline to 13 weeks
Continuous Glucose Monitoring (CGM) measured time with glucose greater than 250 mg/dL | 13 weeks
  Continuous Glucose Monitoring (CGM) measured time with glucose greater than 250 mg/dL from baseline to 13 weeks
Continuous Glucose Monitoring (CGM) measured time with glucose less than 70 mg/dL | 13 weeks
  Continuous Glucose Monitoring (CGM) measured time with glucose less than 70 mg/dL from baseline to 13 weeks
Continuous Glucose Monitoring (CGM) measured time with glucose less than 54 mg/dL | 13 weeks
  Continuous Glucose Monitoring (CGM) measured time with glucose less than 54 mg/dL from baseline to 13 weeks
Continuous Glucose Monitoring (CGM) measured coefficient of variation | 13 weeks
  CGM-measured coefficient of variation from baseline to 13 weeks
Change in glycated hemoglobin (HbA1c) | 13 weeks
  Change in HbA1c from baseline to 13 weeks
Patient Reported Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ), Caregiver | 13 weeks
  Patient-reported outcome (PRO) survey for Insulin Treatment Satisfaction Questionnaire (ITSQ), customized for the study. Inconvenience subscale (items 1-3,15,16; now listed as 1-5) and Delivery System subscale (items 17-22; now listed as 6-11) and one additional item added by study team (#12). Higher scores indicate less treatment satisfaction.
Patient Reported Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ), Participant | 13 weeks
  Patient-reported outcome (PRO) survey for Insulin Treatment Satisfaction Questionnaire (ITSQ), customized for the study. Inconvenience subscale (items 1-3,15,16) and Delivery System subscale (items 17-22). Higher scores indicate less treatment satisfaction.
Patient Reported Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ), Caregiver | 39 weeks
  Patient-reported outcome (PRO) survey for Insulin Treatment Satisfaction Questionnaire (ITSQ), customized for the study. Inconvenience subscale (items 1-3,15,16; now listed as 1-5) and Delivery System subscale (items 17-22; now listed as 6-11) and one additional item added by study team (#12) Higher scores indicate less treatment satisfaction.
Patient Reported Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ), Participant | 39 weeks
  Patient-reported outcome (PRO) survey for Insulin Treatment Satisfaction Questionnaire (ITSQ), customized for the study. Inconvenience subscale (items 1-3,15,16) and Delivery System subscale (items 17-22) Higher scores indicate less treatment satisfaction.
Percentage of participants using Afrezza and basal insulin (Afrezza-BI) regimen | At 13 weeks
  Percentage of participants using Afrezza-BI regimen at time of 13-week visit
Percentage of participants that continue on the Afrezza and basal insulin (Afrezza-BI) regimen | After 13 weeks
  Percentage of participants that continue on Afrezza-BI after 13-week visit
Incidence of Adverse Events of Special Interest (AESIs) | 13 weeks
  Incidence and severity of AESIs which include the following events: acute bronchospasm, clinically relevant decline in pulmonary function (>15% decline from baseline percent predicted FEV1 accompanied by respiratory symptoms), hypersensitivity reactions, including anaphylaxis, hospitalization for asthma, use of corticosteroid bursts for diagnosis of asthma, diagnosis of asthma, diabetic ketoacidosis, severe hypoglycemia
Incidence of Adverse Events of Special Interest (AESIs) | 39 weeks
  Incidence and severity of AESIs which include the following events: acute bronchospasm, clinically relevant decline in pulmonary function (>15% decline from baseline percent predicted FEV1 accompanied by respiratory symptoms), hypersensitivity reactions, including anaphylaxis, hospitalization for asthma, use of corticosteroid bursts for diagnosis of asthma, diagnosis of asthma, diabetic ketoacidosis, severe hypoglycemia
Change in percent predicted FEV1 | 13 weeks
  Change in percent predicted FEV1 from baseline to Week 13
Change in percent predicted FEV1 | 39 weeks
  Change in percent predicted FEV1 from baseline to Week 39
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | 13 weeks
  Incidence and severity of TEAEs and SAEs
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | 39 weeks
  Incidence and severity of TEAEs and SAEs

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Barbara Davis Center for Diabetes Young Adult Clinic, Aurora, Colorado
  - Joslin Diabetes Center, Boston, Massachusetts